CLINICAL TRIAL: NCT01866722
Title: A Test of Two Clinical Methods to Prompt a Quit Attempt Among Smokers
Brief Title: Not Quite Ready to Quit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, John Hughes, Principal Investigator, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHRBS B12-268; R01CA163176 (NIH)
Record Dates: First submitted 2013-05-22; First posted 2013-05-31 (Estimated); Last update posted 2017-07-31 (Actual); Status verified 2017-07

CONDITIONS: Smoking Cessation
Keywords: nicotine dependence; smoking cessation; lapse; relapse; tobacco; quit attempts; abstinence; motivation; reduction
MeSH Terms: conditions — Smoking Cessation; Tobacco Use Disorder; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Usual Care (Active Comparator): Participants will get a brief (<5 min) telephone counseling session about quitting. After that, printed materials with resources to help quitting will be mailed to the participants.
  Interventions: Behavioral: Usual care
- Reduction (Active Comparator): Participants will have 3 telephone counseling sessions that focus on ways to reduce tobacco cigarette smoking. After the final session printed materials with resources to help quitting will be mailed to the participants.
  Interventions: Behavioral: Reduction
- 5Rs (Active Comparator): Participants will have 3 telephone counseling sessions that focus on the 5Rs for quitting tobacco cigarette smoking (Relevance, Risks, Rewards, Roadblocks, Repeat). After the final session printed materials with resources to help quitting will be mailed to the participants.
  Interventions: Behavioral: 5Rs

INTERVENTIONS:
Behavioral: Usual care — Participants will get a brief (<5 min) telephone counseling session about quitting. After that, printed materials with resources to help quitting will be mailed to the participants.
  Arms: Usual Care
Behavioral: Reduction — Participants will have 3 telephone counseling sessions that focus on ways to reduce tobacco cigarette smoking. After the final session printed materials with resources to help quitting will be mailed to the participants.
  Arms: Reduction
Behavioral: 5Rs — Participants will have 3 telephone counseling sessions that focus on the 5Rs for quitting tobacco cigarette smoking (Relevance, Risks, Rewards, Roadblocks, Repeat). After the final session printed materials with resources to help quitting will be mailed to the participants.
  Arms: 5Rs

SUMMARY:
In our communications with the public, the investigators will call this the Not Quite Ready to Quit Smoking Study.

One new method to increase quit attempts is to have smokers reduce their cigs/day. The investigators and others have shown that reduction aided by nicotine medications can increase quit attempts and later abstinence among smokers not ready to quit. Because half of smokers are reluctant to use nicotine medications for a non-cessation reason, the investigators now propose to test whether reduction not aided by nicotine medications can be effective. Another new method to increase quit attempts is motivational counseling. The investigators previously found implementation of the brief United States Public Health Service (USPHS) Guidelines 5 Rs motivational intervention via three 15 min phone calls can provide a large increase in quitting (OR = 6.3); however, the investigators need to replicate that result. A vendor will proactively email adult, daily smokers listed in a consumer panel to recruit 560 smokers who do not plan to quit in the next month and randomize them to a) reduction counseling without the aid of nicotine medications , b) brief counseling guided by the USPHS 5 R's, or c) usual care. The first two conditions will be delivered via brief counseling calls at study onset and then 2 and 4 weeks later (total = 35 min). The usual care condition will consist of a brief (< 5 min) phone intervention followed by a quit guide. Our major hypothesis is that the incidence of quit attempts over the 6 months of the study will be greater in both the reduction and the motivational conditions than in the usual care condition. A secondary hypothesis is that the increase in quit attempts will lead to increased abstinence. Another secondary hypothesis is that beneficial effects of both treatments will be mediated by increases in self-efficacy and intentions to quit. A final hypothesis is that decreases in cigs/day and nicotine dependence will mediate the efficacy of the reduction treatment but not the motivational treatment and, conversely, that a shift in decisional balance will mediate the efficacy of the motivational treatment but not of the reduction treatment.

DETAILED DESCRIPTION:
Objectives

Among smokers who wish to quit at some time but do not plan to quit in the next month:

Major Hypotheses

Major Hypothesis 1: A treatment to reduce cigs/day that does not include nicotine replacement therapy (NRT) will increase the incidence of a quit attempt (yes/no outcome).

Major Hypothesis 2: A motivational treatment based on the USPHS's 5 Rs will increase the incidence of a quit attempt (yes/no outcome)

A comparison of the two active conditions is not an objective of the study.

The current application focuses on new clinical interventions to increase quit attempts. One recent method to increase quit attempts in ambivalent smokers has been reduction of cigs/day. This method typically includes teaching ways to reduce cigs/day with the aid of nicotine replacement therapy (NRT). Recent reviews and meta-analyses have concluded reduction aided by NRT among ambivalent smokers consistently increases the probability of future quit attempts and abstinence.

Another recent clinical method to prompt quit attempts is motivational treatments. The USPHS treatment guidelines recommend smokers not ready to quit receive a briefer, somewhat different motivational treatment focusing on the "5 Rs;" i.e., a) personal relevance of smoking, b) risks of smoking, d) rewards from smoking cessation, d) roadblocks to quitting and e) repetition.

Rationale for Proposed Studies: We now propose to test the efficacy of a non-pharmacological reduction treatment for two reasons. First, many smokers are not willing to use NRT for reduction. Another reason for testing a non-pharmacological treatment for reduction is that prior studies of NRT- aided reduction have been interpreted to indicate that reducing cigs/day will increase later quitting; however, since many(but not all)recent studies suggest pretreatment with NRT alone improves quitting, it is unclear whether reduction or pretreatment is the cause of any increase quitting in prior studies.

We also propose a replication test of our 5 Rs intervention because, although the counseling technique of reviewing Relevance, Risks, Rewards, Roadblocks, and Repeat (5R's) have been part of the last two USPHS Guidelines (most recently updated in 2008), our search of PubMed, PsychINFO, NIH RePorter (database of NIH grants) and clinicaltrials.gov in 11/11 indicates no published and no current or planned test of the 5 Rs, other than our study (Carpenter et al., 2004). Clearly, more than one test of the approach recommended for >80% of smokers who are not ready to quit (Wewers, Stillman, Hartman, & Shopland, 2003) is needed. Another reason for our replication test is that our prior Journal of Consulting and Clinical Psychology (JCCP) study of the 5 Rs used a no treatment control group; thus, we wish to increase clinical relevance and methodological rigor by employing a usual care comparison condition.

Study Design Design and Rationale for Methodological Decisions: We will use a three-group (n= 560 total)Randomized Control Trial (RCT) to test whether a reduction and a 5 Rs motivational intervention each increases the incidence of a quit attempt (Table 2). The reduction and 5 Rs interventions will be time-matched with an initial 15 min call at baseline followed by two 10 min calls at 2 and 4 weeks later (total = 35 min). The usual care condition will receive a brief (< 5 min) call and mailed information about risks of smoking, self-quitting and treatment resources at the same time-points. Monitoring of cigs/day and abstinence will be via weekly online questionnaires.

Timing of treatments and measure Counseling calls Usual care: at baseline only Reduction: baseline, Week 2, Week 4 5Rs: baseline, Week 2, Week 4

Measures for all 3 groups--all asked weekly x 4 then monthly x 5 cigs/day quit attempts abstinence mediators Subject Selection Subjects will be current smokers who do not plan to quit in the near future; i.e., about 70% of all smokers, because the purpose of our treatment is to prompt new quit attempts among ambivalent smokers.

Vulnerable Populations Not applicable

Number of Subjects 560 current smokers. We will consent 560 in an effort to have 516 who complete at least one counselor call.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* smoke > 10 cigs/day seven days/week,
* wants to stop at some point but have no plans to quit in the next month
* is able to read and write English
* is a US citizen or a permanent resident alien
* available for counseling calls before 20:00 Eastern Time

Exclusion Criteria:

* has reduced cigs/day by > 25% in the last month
* has used non-cigarette tobacco in the last month
* has used electronic cigarettes, nicotine replacement medications, varenicline or bupropion in the last month

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 560 (Estimated)
Dates: Start 2013-09 (Actual); Primary Completion 2015-01-10 (Actual); Study Completion 2015-07-14 (Actual)

PRIMARY OUTCOMES:
quit attempts | About 2 years
  The incidence of an attempt to quit smoking tobacco cigarettes during the 6 months of the study.

SECONDARY OUTCOMES:
abstinence | About 2 years
  7 day point prevalence abstinence from smoking tobacco cigarettes at 6 months after the beginning of treatment.

OTHER OUTCOMES:
prolonged abstinence | about 2 years
  Abstinence from tobacco cigarette smoking during the last 3 months of the study

CONTACTS AND LOCATIONS:
Overall Officials: John R Hughes, MD, Principal Investigator — University of Vermont
Locations (1):
- University of Vermont, Burlington, Vermont, United States

REFERENCES:
- [Background] Wewers ME, Stillman FA, Hartman AM, Shopland DR. Distribution of daily smokers by stage of change: Current Population Survey results. Prev Med. 2003 Jun;36(6):710-20. doi: 10.1016/s0091-7435(03)00044-6. PMID 12744915
- [Background] Carpenter MJ, Hughes JR, Keely JP. Effect of smoking reduction on later cessation: a pilot experimental study. Nicotine Tob Res. 2003 Apr;5(2):155-62. doi: 10.1080/146222003100007385. PMID 12745487
- [Result] Klemperer EM, Hughes JR, Solomon LJ, Callas PW, Fingar JR. Motivational, reduction and usual care interventions for smokers who are not ready to quit: a randomized controlled trial. Addiction. 2017 Jan;112(1):146-155. doi: 10.1111/add.13594. Epub 2016 Oct 5. PMID 27566993